CLINICAL TRIAL: NCT00277199
Title: Study to Compare the Pharmacokinetics of CD-CHO1 Process BMS-188667 to DE Process BMS188667 in Healthy Subjects
Brief Title: Comparability DE vs CD-CHO1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-017; 016149
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Abatacept

INTERVENTIONS:
Drug: Abatacept

SUMMARY:
Study to Compare the Pharmacokinetics of CD-CHO1 Process BMS-188667 to DE Process BMS-188667 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Healthy subjects as determined by good health as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs and clinical laboratory determinations.
* Body weight for all subjects will be <- 100 kg.
* body Mass Index (BMI) of 18-30 kg/m2 inclusive; BMI = weight (kg)/[height (m)]2
* Men and women (not nursing, not prgnant), who are at least 18 years of age. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study for at least 4 weeks before and for up to 10 weeks after the infusion of BMS-188667 in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* WOCBP and males who are unwilling or unable to use an acceptable method to avoid pregnancy for up to 10 weeks after he infusion of BMS-1886678. WOCBP must also be using an acceptable method of contraception for at least 1 month before dosing.
* Women who are pregnant ore breast-feeding.
* Women with positive pregnanacy tes on enrollment or prior to study drug administration.
* History or current evidence of any signiicant acute or chroinic medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
To test pharmacokinetics

SECONDARY OUTCOMES:
To test Safety and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Inveresk Clinical Research, Edinburgh, United Kingdom